CLINICAL TRIAL: NCT00527696
Title: Randomized Clinical Trial Comparing TVT SECUR System (TVT S) and Trans Vaginal Obturator Tape (TVT-O) for Surgical Management of Stress Urinary Incontinence
Brief Title: Trial Comparing TVT SECUR System and Trans Vaginal Obturator Tape for Surgical Management of Stress Urinary Incontinence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: statistical Significance was reached for primary outcome
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ken Maslow, Assistant professor, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B2007:044
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TVT SECURE (Active Comparator): sling
  Interventions: Procedure: transvaginal obturator tape
- TVT O (Active Comparator): sling
  Interventions: Procedure: transvaginal obturator tape

INTERVENTIONS:
Procedure: transvaginal obturator tape

SUMMARY:
To compare the efficacy and complications of the TVT SECUR system (TVT S) and trans-vaginal obturator tape (TVT-O) procedures for the surgical management of female stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with symptoms of stress urinary incontinence and a positive cough test who require surgical management. Cough test is positive when leakage of urine is seen from the urethra synchronously with the patient performing a cough or valsalva manuver with a comfortably full bladder in the lying or standing position.

Exclusion Criteria:

* Women with predominantly symptoms of urge urinary incontinence
* Presence of prolapse greater than Pelvic organ prolapse quantification (POPQ) Stage 1 or prolapse requiring surgery
* Detrusor overactivity on cystometrogram at urodynamic testing
* Previous surgery for incontinence
* Intrinsic sphincter deficiency (MUCP<20 cm H2O or Q -tip <30o)
* Voiding dysfunction with postvoid residual >100 cc

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Objective cure as defined by the cough test at one year from surgery | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ken D Maslow, MD, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839
- [Derived] Maslow K, Gupta C, Klippenstein P, Girouard L. Randomized clinical trial comparing TVT Secur system and trans vaginal obturator tape for the surgical management of stress urinary incontinence. Int Urogynecol J. 2014 Jul;25(7):909-14. doi: 10.1007/s00192-013-2312-7. Epub 2014 Jan 23. PMID 24452619